CLINICAL TRIAL: NCT00724490
Title: Unilateral Deep Brain Stimulation of the Nucleus Accumbens in Patients With Treatment Resistant Obsessive Compulsive Disorder
Brief Title: Unilateral Deep Brain Stimulation (DBS) of the Nucleus (Nucl.) Accumbens (Acc.) in Patients With Treatment Resistant Obsessive Compulsive Disorder (OCD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Joachim Klosterkoetter, MD, Department of Psychiatry, University of Cologne, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ocdbs-Psy-120304
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2008-07-29 (Estimated); Status verified 2008-07

CONDITIONS: Obsessive Compulsive Disorder
Keywords: Deep Brain Stimulation; Obsessive Compulsive Disorder; Nucleus Accumbens
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Deep Brain Stimulation — Unilateral Deep Brain Stimulation in the right Nucleus Accumbens
  Other Names: Model 3387 DBS Lead, Medtronic, Minneapolis, USA

SUMMARY:
The purpose of the study was to evaluate whether a unilateral Deep Brain Stimulation of the right Nucleus Accumbens could lead to a more than 35% reduction of symptoms in patients with a treatment resistant Obsessive Compulsive Disorder within two years.

DETAILED DESCRIPTION:
From the late ninety's on, a few work groups published the case series of patients with treatment resistant OCD undergoing deep brain stimulation (DBS). This stereotactical method involves surgically implanted electrodes and previously has been used primarily for the treatment of Parkinson's disease and tremor.

In almost all reported cases, a bilateral stimulation in the anterior limb of the internal capsule (ALIC was applied. However, the electrode designs between the groups varied and in some cases the stimulation area was extended to the adjacent ventral striatal regions including the nucleus accumbens (NAC).

Cortical-striate-thalami-cortical (CSTC) circuits are supported to be implicated in the pathogenesis underlying OCD caused by a failure of inhibition of the ventral striatum. Together with other structures the nucleus accumbens forms the ventral striatum. Because of the predominant role of the NAC to exert modulatory effects within these circuits we considered it to provide a promising target location for DBS.

Moreover the NAC ventrally borders with the anterior limb of the internal capsule and the subventricular lateral fundus of the nucleus accumbens is even permeated in rostral sections by numerous internal capsule fiber bundles. It was therefore to be expected that the electrode trajectories and stimulation target selected by us additionally would have an effect on the fibre systems of the internal capsule.

The NAC had been introduced as primary target for DBS in treatment resistant OCD by our group. Pilot series showed that the right stimulation of the NAC yielded the best results, whereas bilateral stimulation showed no additional benefit.

ELIGIBILITY:
Inclusion Criteria:

* Obsessive compulsive disorder (according to DSM IV-criteria) as the primary psychiatric diagnosis
* severity level of OCD more than 25 on the Yale-Brown Obsessive Compulsive Scale
* course of illness had to have been present for at least five years in a chronic or progressive form despite any treatment trials (treatment resistance)
* treatment resistance: at least two serotonin reuptake inhibitors (SSRI´s), or one SSRI and clomipramine in sufficient dosages for at least 10 weeks, an augmentation trial with lithium, buspirone or a neuroleptic lasting at least 10 weeks, and complete cognitive-behavioral psychotherapy, including "exposure and response prevention" of a minimum of 20 sessions with a documented lack of efficiency
* the ability to give written and informed consent

Exclusion Criteria:

* co-morbid psychotic disorder according to DSM-IV criteria
* suicidal tendencies in the last 6 months
* history of cerebral trauma
* clinically relevant internal or neurological disorder
* substance misuse or dependence in the last six months
* ineligibility to fulfill the neurosurgical and anesthesiological preconditions for the implantation of a DBS
* pregnancy
* lactation period

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2004-02; Primary Completion 2007-09 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale | Baseline (preoperative), 1week, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months

SECONDARY OUTCOMES:
Beck Depression Inventory | Baseline (preoperative), 1 week, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Klosterkötter, MD, Principal Investigator — Department of Psychiatry, Head of Department, University of Cologne
Locations (1):
- Department of Psychiatry, University of Cologne, Cologne, North Rhine-Westphalia, Germany